CLINICAL TRIAL: NCT00205907
Title: Phase 1/Phase 2 Study of the Aeris Bronchoscopic Lung Volume Reduction (BLVR) System in Patients With Advanced Emphysema
Brief Title: Israeli 10 mL Bronchoscopic Lung Volume Reduction (BLVR) Phase 1/2 Emphysema Study - Initial Formulation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in Formulation
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Edward P Ingenito, MD, PhD, Medical Director & CSO, Aeris Therapeutics Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C04-003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-02

CONDITIONS: Pulmonary Emphysema
Keywords: BLVR; emphysema; COPD; COLD; chronic obstructive pulmonary disease; pulmonary emphysema
MeSH Terms: conditions — Pulmonary Emphysema; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single (Experimental): BLVR treatment
  Interventions: Biological: BLVR Hydrogel

INTERVENTIONS:
Biological: BLVR Hydrogel — 10 mL BLVR Hydrogel

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Aeris BLVR System in patients with advanced emphysema.

DETAILED DESCRIPTION:
Emphysema is a progressive, debilitating disease that affects nearly 3 million people in the United States or roughly one percent of the US population. The disease is characterized by destruction of lung tissue as a result of inflammation caused by exposure to noxious inhaled agents for extended periods. The most common cause of this condition is cigarette smoking, although genetic and occupational causes account for up to 10% of cases. Despite aggressive public health initiatives aimed at discouraging the use of cigarettes, smoking-related lung diseases remain a significant cause of disability and death in the United States. Currently there are 46 million smokers in the US. Due to the number of current and new smokers, emphysema is expected to remain a leading cause of morbidity and mortality in the United States for years to come.

Aeris has developed a novel bronchoscopic system for achieving the benefits of lung volume reduction without surgery. The Bronchoscopic Lung Volume Reduction (BLVR) Hydrogel System, a new investigational therapy for emphysema, is intended to reduce lung volume over a period of weeks by collapsing and promoting the remodeling of diseased areas of the lung. The resulting reduction in lung volume is intended to restore a more normal physiological relationship between lung and chest wall, improve breathing and exercise capacity and alleviate symptoms of chronic dyspnea. The current study will evaluate the safety and efficacy of this procedure in patients with advanced emphysema.

ELIGIBILITY:
Inclusion Criteria include:

* Clinical diagnosis of advanced heterogeneous emphysema
* Age > 18 years at the time of initial presentation
* Clinically significant dyspnea (MRC Dyspnea >/= 2)
* Failure of standard medical therapy to provide relief of symptoms
* BUN, creatinine, ALT, AST, alkaline phosphatase, WBC, hematocrit, platelet count, PT and PTT within normal limits
* Pulmonary function tests

Exclusion Criteria:

* Alpha-1 protease inhibitor deficiency verified by a serum level of < 80 mg% or knowledge of PI*ZZ genotype
* Body mass index < 15 kg/m2 or > 35 kg/m2
* Clinically significant asthma (reversible airway obstruction), chronic bronchitis or bronchiectasis
* Tobacco use within 16 weeks of the initial clinic visit
* Allergy to fish or pork products or sensitivity to tetracycline
* FEV1 <20% with DLCO <20% or homogeneous disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-01; Primary Completion 2006-08 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Product-related life-threatening adverse events, permanently disabling complications and deaths | 1 year post treatment
FEV1 | 12 weeks post treatment
MRC Dyspnea Score | 12 weeks post treatment
Six-Minute Walk Test | 12 weeks post treatment
Health-Related Quality of Life | 12 weeks post treatment

SECONDARY OUTCOMES:
Lung function tests | 12 weeks post treatment
Lung volume measures | 12 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Issahar Ben-Dov, MD, Principal Investigator — The Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba (Tel Hashomer) Medical Center, Ramat Gan, Israel

REFERENCES:
- See also: Ingenito EP, Berger RL, Henderson AC, Reilly JJ, Tsai L, Hoffman A. Bronchoscopic lung volume reduction using tissue engineering principles. Am J Respir Crit Care Med. 2003 Mar 1;167(5):771-8. Epub 2002 Oct 11. — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi